CLINICAL TRIAL: NCT07002567
Title: Predictors of Motor İmagery Performance in Cerebral Palsy
Status: Not yet recruiting | Type: Observational
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Seda AYAZ TAŞ, Assistant Professor, Abant Izzet Baysal University
Other Study IDs: BAIBU-FTR-SAT-11
Record Dates: First submitted 2025-05-24; First posted 2025-06-03 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-05

CONDITIONS: Cerebral Palsy (CP); Spasticity; Motor Learning
Keywords: MOTOR İMAGERY; CEREBRAL PALSY; UPPER EXTREMİTY; PHYSIOTHERAPY
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Unilateral cerebral palsy: Cerebral Palsy (CP) is a group of permanent disorders in activity limitation, motor and posture development due to non-progressive damage to the developing fetus or infant brain. In spastic unilateral CP, involvement occurs unilaterally in one half of the body.
  Interventions: Other: Implicit motor imagery; Other: Explicit motor imagery
- Bilateral cerebral palsy: Cerebral Palsy (CP) is a group of permanent disorders in activity limitation, motor and posture development due to non-progressive damage to the developing fetus or infant brain. In spastic bilateral CP, involvement is seen bilaterally in all 4 extremities.
  Interventions: Other: Implicit motor imagery; Other: Explicit motor imagery

INTERVENTIONS:
Other: Implicit motor imagery — Implicit motor imagery is the ability to engage with the projection and manipulation of the body schema from a first-person perspective. Implicit motor imagery skills were evaluated Recognize App Recognize Hand Hand Laterality Task with, developed by NOI group. (http://www.noigroup.com/ Recognise).
Other: Explicit motor imagery — In explicit motor imagery, the person simulates a specific motor movement, that is, the individual is aware that she is imagining the movement.Explicit motor imagery skills were evaluated with Movement Imagery Questionnaire for Children (MIQ-C), mental chronometry and box block test.

SUMMARY:
There are very few studies in the literature examining the effect of age on motor imagery ability in children with cerebral palsy. To our knowledge, no studies have investigated the impact of other related factors. The aim of this study is to investigate the effects of age, sex, body mass index, Gross Motor Function Classification System (GMFCS) level, and Manual Ability Classification System (MACS) level on motor imagery abilities in children with cerebral palsy.

H1-1: Age has an effect on motor imagery abilities in children with cerebral palsy.

H1-2: Sex has an effect on motor imagery abilities in children with cerebral palsy.

H1-3: Clinical type has an effect on motor imagery abilities in children with cerebral palsy.

H1-4: Body mass index has an effect on motor imagery abilities in children with cerebral palsy.

H1-5: GMFCS level has an effect on motor imagery abilities in children with cerebral palsy.

H1-6: MACS level has an effect on motor imagery abilities in children with cerebral palsy.

DETAILED DESCRIPTION:
Cerebral Palsy (CP) is a group of permanent movement and posture disorders resulting from non-progressive damage to the developing brain. Along with motor impairments, individuals with CP often experience sensory, cognitive, communication, behavioral, and musculoskeletal challenges. The most widely accepted classification, developed by the Surveillance of Cerebral Palsy in Europe (SCPE), categorizes CP into spastic, dyskinetic, and ataxic types. Spastic CP is the most common and may present with either bilateral or unilateral involvement. Dyskinetic CP includes dystonic and choreoathetotic subtypes.

Motor learning involves acquiring new skills to improve movement quality. While typically developing children learn motor activities naturally, children with CP may experience difficulties due to structural and motor planning deficits. Motor imagery (MI), defined as mentally simulating a movement without physical execution, is one strategy that supports motor learning. MI and actual movement engage similar brain regions and share cognitive and neurophysiological components.

MI can be experienced from a visual or kinesthetic perspective. Visual imagery involves watching the movement as an observer, while kinesthetic imagery involves internally experiencing the movement as the actor. Kinesthetic imagery is more closely associated with motor planning and functional improvement. MI can be explicit, involving conscious simulation of movement, or implicit, occurring unconsciously through internal body representations. Both forms are used in neurorehabilitation.

Previous studies on MI in children with CP have typically included participants aged 6 to 20 with relatively good motor and functional abilities. Although some researchers suggest that MI skills begin to develop between the ages of 5 and 7, findings are inconsistent, highlighting the need for further investigation.

Research exploring factors that may influence MI ability in children with CP is limited. While age has been studied to a small extent, the effects of sex, clinical type, body mass index (BMI), Gross Motor Function Classification System (GMFCS) level, and Manual Ability Classification System (MACS) level have not been thoroughly examined. This study aims to explore the influence of these variables on MI ability in children with CP. After recording the children's demographic characteristics (age, sex, height, weight, body mass index [BMI], and duration of physiotherapy), the following assessments will be conducted:

Gross Motor Function Classification System (GMFCS):

GMFCS is a five-level classification system used to assess gross motor function in individuals with CP, focusing on sitting, transfers, and mobility. It categorizes function based on self-initiated movement across specific age bands: 0-2, 2-4, 4-6, 6-12, and 12-18 years. Level I indicates independent walking with minimal limitations, while Level V indicates the need for a wheelchair for mobility.

Manual Ability Classification System (MACS):

MACS is used to classify how children with CP (aged 4-18 years) use their hands to handle objects in daily life. Level I indicates the highest manual ability, with ease in handling objects, while Level V indicates very limited ability and the need for maximum assistance.

Hand Laterality Task:

Implicit motor imagery ability will be assessed using the Hand Laterality Task, which requires participants to identify whether an image shows a left or right hand. The Recognise Hand app, developed by the NOI group, will be used for this purpose. Outcome measures include response accuracy (percentage of correct responses) and reaction time.

Mental Chronometry Task:

Explicit motor imagery will be assessed using the mental chronometry paradigm. Participants will first perform a physical movement and then imagine performing the same movement toward targets at varying distances. The duration of the actual and imagined movements will be recorded. The Box and Block Test will be used, and temporal congruence will be calculated using the delta time formula: [(actual movement time - imagined movement time) / ((actual movement time + imagined movement time) / 2)] x 100.

Box and Block Test:

This test evaluates manual dexterity and is commonly used in both clinical and research settings due to its simplicity and cost-effectiveness. Participants are instructed to move as many blocks as possible from one compartment to another in 60 seconds. The score reflects the number of successfully transferred blocks, with higher scores indicating better upper extremity performance. It will also be used in the mental chronometry task.

Movement Imagery Questionnaire for Children:

This questionnaire evaluates visual (internal, external) and kinesthetic imagery abilities. It includes 12 items: 4 for each imagery type. Participants will perform four movements physically and then imagine them from each perspective. Imagery vividness will be rated on a 7-point Likert scale (1 = very hard to feel, 7 = very easy to feel). Higher scores indicate better imagery ability.

ELIGIBILITY:
Inclusion Criteria:

* 6-18 year olds diagnosed with spastic type unilateral and bilateral diplegia CP,
* Those with Gross Motor Function Classification System (GMFCS) level I - II,
* Hand Skill Classification System (EBSS) level I-II,
* Children with a Mini-Mental Test score of at least 24 points,
* Those with IQ <70, Those who can understand the guidelines of the study

Exclusion Criteria:

* Those with advanced vision, hearing and attention problems,
* Those with advanced cardiovascular or cognitive problems,
* Upper extremity botulinum toxin administration and surgery in the last 6 months,
* Those who have received MI training in the last 6 months

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: This study included between the ages 6 and 18 years 27 children with unilateral and 27 bilateral cerebral palsy with level 1 or 2 according to the Gross Motor Function Classification System (GMFCS), Manual Ability Classification System (MACS),
Sampling Method: Non-Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2025-07-04 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Explicit motor imagery -1 | 2 years
  Box and block test,Participants were first asked to pass the maximum number of wooden blocks to the other side of the wooden box in 60 seconds, three times for each hand. The actual number of movement blocks was obtained by calculating the average of 3 applications. Then, each participant was asked to visually pass the maximum number of wooden blocks to the other side of the wooden box without moving, three times for both hands. While visualizing, the participants pressed the button in front of them for each wooden block they placed, thus the number of wooden blocks they imagined passing to the other side was seen. The number of imaged movement blocks was obtained by taking the average of 3 applications. The number of wooden blocks passed with actual movement and imagined movement was compared.

SECONDARY OUTCOMES:
Explicit motor imagery - 2 | 2 years
  Box and block test, mental chronometry, The mental chronometry paradigm was evaluated using the wooden box and 10 wooden blocks of the box block test. The participants were first asked to grasp 10 wooden blocks from one side of the wooden box and pass them to the other side, three times in both hands, and the time taken was calculated with a stopwatch. Then, they were asked to visualize passing 10 wooden blocks to the other side of the wooden box, 3 times for each hand, and to say when they imagined that all 10 wooden blocks had passed. When they said they were done, the stopwatch was stopped. The application was performed three times on the dominant and non-dominant sides for real and imagined movements, and the average was noted. Delta time was calculated based on real and imagined movement time. . Delta time is calculated with the formula =[(real movement-imagined movement) / [(real movement+imagined movement) / 2]x100.
Explicit motor imagery - 3 | 2 years
  Movement Imagery Questionnaire for Children (MIQ-C),The Movement Imagination Questionnaire for Children will be used to measure visual (intrinsic, extrinsic) and kinesthetic imagery ability. It contains a total of 12 items: 4 items on internal, 4 items on external, and 4 items on kinesthetic visualization skills. Within the scope of the survey, the individual will be asked to visualize 4 different movements from 3 different visualization perspectives. The individual will be expected to first actually perform the movement in the instruction once and then imagine doing the movement. The clarity of this imagery will be rated using a Likert-type scale from 1 (very difficult to feel) to 7 (very easy to feel). A higher score from the test indicates higher imagination ability.
Implicit motor imagery | 2 years
  Hand Laterality Task, Implicit motor imagery capacity was assessed with the Laterality Task (choice task). Laterality task is based on deciding which side of the photograph belongs to the limb shown. Recognize Hand is an application developed by the NOI group and used to evaluate right-left discrimination.(http://www.noigroup.com/ Recognise). In terms of imagination ability and hand laterality, the sharpness of the choices made in right-left discrimination (percentage of correct answers) and the reaction time during the choice were evaluated.

CONTACTS AND LOCATIONS:
Locations (3):
- Turkey (Türkiye) (3):
  - Kdz. Ereğli Gökkuşağı Özel Eğitim ve Rehabilitasyon Merkezi, Zonguldak, Ereğli
  - Bolu Abant İzzet Baysal University, Bolu, Gölköy
  - Düzce Gökkuşağı Özel Eğitim ve Rehabilitasyon Merkezi, Düzce, Merkez

IPD SHARING:
Plan to Share IPD: No